CLINICAL TRIAL: NCT01598519
Title: School-based Comprehensive Suicide Intervention in Shanghai, China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Pu Dong Institute of Education Development (Unknown); Shanghai Sanling North Junior Middle School (Unknown); Shanghai Shangnan East Junior Middle School (Unknown); Shanghai Sanling Senior Middle School (Unknown); Shanghai Yangsi Senior Middle School (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007BAI17B03
Record Dates: First submitted 2012-02-06; First posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Suicide
Keywords: school-based; adolescent suicide; intervention; screening
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (Experimental): 1500 students are randomized to receive a universal suicide intervention apart from usual school psychology classes. Furthermore, high risk of suicidal students screened in study group will receive an indicated suicide intervention in addition to usual school psychology classes.
  Interventions: Behavioral: suicide intervention
- control group (No Intervention): 1500 students are randomized to receive usual school psychology classes. High risk of suicidal students screened in control group will receive usual psychology classes.

INTERVENTIONS:
Behavioral: suicide intervention — universal intervention:(1)students: 4 sections about cherishing life, coping strategies, suicide and depression disorder during 2 semesters, each session lasting 45 minutes.(2)gatekeeper: 4 sessions about teenagers psychological crisis intervention strategies during 2 semesters, 30minutes per session.
  indicated intervention: (1)student: 2 semesters, 20 sessions' group life skill and cognitive-behavioral psychological training lesson, including Youth rational emotive group tutoring(eight classroom sessions), Coping skill group tutoring(six classroom sessions)and Behavior group tutoring(six classroom sessions), once a week, each session lasting 1.5hours.(2)gatekeeper: a social support net.
  Arms: study group

SUMMARY:
The primary aim of this study is to examine whether a school-based suicide intervention is effective in reducing suicide related risk factors in a population of middle and high students. It hypothesized that receiving the intervention will reduce the severity of suicide related risk factors such as depression, hopelessness, suicidal behaviors and increasing protective factors such as social support, self esteem, suicide knowledge and attitude and so on, as compared to the control group.

DETAILED DESCRIPTION:
A total of 3000 students from two junior schools (grade 7 and 8) and two senior schools (grade 10 and 11) in Shanghai Pu Dong district were recruited in our study. All students were randomly assigned into universal study group or universal control group by class level. In those two groups, high risk of suicidal students were identified by screening. A universal suicide intervention was conducted in the universal study group; an indicated suicide intervention was conducted in the indicated study group. All students in universal study group and universal control group completed the self-administered questionnaire before and 6 months after the end of universal intervention. High risk of suicidal students in the indicated study group and indicated control group completed another self-administered questionnaire before, 6 months and 18 months after the end of the indicated intervention.

ELIGIBILITY:
Inclusion Criteria:

* students of grade 6,7,9,10 from four schools (2 middle schools, 2 high schools)

Exclusion Criteria:

* students who are not attending school because of long term sickness or moving to other school,or going aboard, etc.
* students whose parents don't agree to participate the study

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
students' score of mediating factors and suicide behaviors | "Change from baseline in suicide behavior at 6 months after the end of the intervention" and "Change from baseline in suicide behavior at 18 months after the end of intervention"

SECONDARY OUTCOMES:
students' score of suicide knowledge and attitude | "Change from baseline in suicide knowledge at 6 months after the end of the intervention" and "Change from baseline in suicide knowledge at 18 months after the end of intervention"

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China